CLINICAL TRIAL: NCT02832193
Title: Retrospective Evaluation of POCD Data of Studies From the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK) Charité - Universitätsmedizin Berlin
Brief Title: Retrospective Evaluation of POCD Data of Studies From KAI, Charité - Universitätsmedizin Berlin
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charite University, Berlin, Germany
Other Study IDs: POCD-Registry
Record Dates: First submitted 2016-06-28; First posted 2016-07-14 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group: POCD data of study patients of the following studies:
  Phydelio - Eudract.-No.: 2008-007237-47 - 08/0618 ZS EK11 Neuprodex - Eudract-No.: 2013 -000823-15 - 13/0491 ZSEK11 BioCog - EA2/092/14 Cognitive Outcome after two stage liver operation - EA1/296/12 ReCosa - EA1/056/13 Hypnoc - EA1/273/11 Sudoco - EA1/242/08 Peratecs - EA1/241/08 Hipster - Eudract.-No.: 2009-016043-19 100/10 ZS EK15 Pain-Long-EA2/041/17 PCI - EA2/024/18 PODSPA - EA4/138/18, PRÄP-GO -EA1/225/19, ANA-PRÄP-Go (EA1/266/20) Further studies from the Department of Anesthesiology and Operative Intensive Care Medince (CCM/CVK), Charité - Universitätsmedizin Berlin
- Control group I: POCD data of prospective control subjects/patients (ASA I+II+III) and POCD data of control subjects/patients of the following studies:
  Neuprodex - Eudract-No.: 2013 -000823-15 - 13/0491 ZSEK11 Phydeliostudie - Eudract.-No.: 2008-007237-47 - 08/0618 ZS EK11 BioCog - EA2/092/14 Cognitive Outcome after two stage liver operation - EA1/296/12 Hypnoc - EA1/273/11 Sudoco - EA1/242/08 Peratecs - EA1/241/08 Hipster - Eudract.-No.: 2009-016043-19 100/10 ZS EK15 BioCog-Studie - EA2/092/14 REACT-Studie - EA2/091/15 PAINLONG-Studie - EA2/041/17 PCI - EA2/024/18 PODSPA - EA4/138/18, PRÄP-GO -EA1/225/19, ANA-PRÄP-Go (EA1/266/20) Further studies from the Department of Anesthesiology and Operative Intensive Care Medince (CCM/CVK), Charité - Universitätsmedizin Berlin

SUMMARY:
Data on prevention of perioperative neurocognitive disorders (pNCDs) are limited. The purpose of this monocentric parallel - grouped observational registry is to collect study data from studies with pNCDs as primary or secondary endpoint to estimate prevalence and incidence of pNCDs.

DETAILED DESCRIPTION:
Perioperative cognitive trajectories (Perioperative neurocognitive disorders [pNCDs]) are described with formal cognitive testing (neurocognitive test battery). Definitions are based on current nomenclature recommendations (Evered et al.) according to DSM-V criteria including a multi-component cognitive test battery comparing baseline and postoperative follow-up testing of patients with cognitive test performance of non-surgical control groups.Cognitive concern and functional ability are described with items from questionnaires, e.g. IQCODE, MMQ, GDS, ADL/IADL and others specific to the respective study design.

Repeated cognitive testing with a battery of computerized neuropsychological tests (Cambridge Neuropsychological Test Automated Battery [CANTAB®]) and non computerized (paper based)tests (e.g. trailmaking test, Grooved pegboard test, Stroop color word interference test, animal naming test, etc.) are performed at preoperative baseline, after 5-7 days and at three months follow up, 1 year, 2 years and 5 years follow-up according to the study design of the registered studies.

Different calculation methods will be applied to the cognitive test data, primarily the dichotomousapproach established by Rasmussen et al. in the International Study on postoperative cognitive deficits (ISPOCD). This calculation method defines POCD as a reliable change in pre- and postoperative cognitive performance (difference scores) of each individual in the surgical patients cohort as compared to the changes in a non-surgical control group (reliable change index in either a composite score including cognitive test parameters from all tests in the cognitive test battery or in at least two of the chosen cognitive test parameters). Additional calculation methods like "g-factor", "GCP" and arbitrary definitions e.g. "20.20- rule" will be used for detailed methodologic evaluation.

In two subprojects we plan to describe domain-specific changes in formal cognitive testing over the registered surgical cohorts.

Subproject 1-Analyses will be performed in joint evaluation with Monument Therapeutics (Spin off Cambridge Cognition). The analyses aim to :

1. Describe cognitive change based on raw cognitive data from the applied cognitive test battery (computerized tests with CANTAB eclipse, CANTAB research suite, CANTAB connect and non-computerized tests)
2. Identify predisposing factors (e.g. patient characteristics, biomarkers, medications) predictive of cognitive decline following surgery
3. Identify the cognitive domains most sensitive to neuropsychological change following surgery

Subproject 2-Analyses will be performed in joint evaluation with Cambridge Cognition. The analyses aim to :

Facilitate the use of data collected from non-surgical controls as normative material for future studies in the research area.

ELIGIBILITY:
Study Group

Inclusion Criteria:

* Age 18 -100 years
* Male or female patients undergoing elective surgery expected to last at least 60 min, screened at the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany
* Written informed consent to participate after having been properly instructed

Exclusion Criteria:

* Lacking willingness to take part in the study, or to have relevant study data collected, saved and analyzed for the purpose of the study
* Accommodation in an institution due to an official or judicial order
* Insufficient knowledge of German language
* Members of the hospital staff
* Homelessness or other conditions that disable reachability for postoperative assessment by post or telephone
* Illiteracy
* Patients who had a history of neurologic deficits (e.g. stroke, history of seizures, etc.)
* Hearing impairment that severely affects the neuropsychological testing.
* Visual impairment that severely affects the neuropsychological testing.
* Participation in other prospective clinical interventional trials

Control Group

Inclusion Criteria:

* Age 18 - 100 years
* Male or female patients (ASA Status I, II+III)
* No planned surgery during the next 3 months
* No surgery during the past 6 months before study inclusion
* Written informed consent to participate after having been properly instructed

Exclusion Criteria:

* Insufficient knowledge of German language Lacking willingness to take part in the study, or to have relevant study data collected, saved and analyzed for the purpose of the study
* Neuropsychiatric conditions that severely affect the neuropsychological testing
* Hearing impairment that severely affects the neuropsychological testing
* Visual impairment that severely affects the neuropsychological testing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients undergoing surgery, screened at the Department of Anesthesiology and Operative Intensive Care Medicine (CCM, CVK), Charité - Universitätsmedizin Berlin, Berlin, Germany
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2009-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive Disorder (NCD) | Up to 1 year
  Mild / major neurocognitive disorder 3 (mild / major NCD 'Postoperative cognitive dysfunction (POCD)') and 12 months (mild / major NCD) postoperatively.
Postoperative cognitive dysfunction (POCD) | Up to 1 year
  Postoperative cognitive dysfunction (POCD) is defined as relevant change in postoperative cognitive performance compared to baseline (preoperative) cognitive performance.

SECONDARY OUTCOMES:
Suspected neurocognitive disorder due to MiniCog | Up to 5 years
  The MiniCog is used for cognitive screening. A cut-off value of <3 points is interpreted possible mild / major NCD. The Mini-Cog consists of a sub-test for word memory skills and a clock drawing test.
Suspected dementia from MOCA | Up to 5 years
  The Montreal Cognitive Assessment (MOCA) with cut-offs according to normative age-adjusted values is used as dementia screening. The MOCA consists of 13 items, which are rated on a scale from 0 to 30 points.
Neurocognitive Disorder (NCD) | Up to 5 years
  Mild / major neurocognitive disorder (mild / major NCD) 60months postoperatively.
Suspected postoperative neurocognitive disorder (mild / major NCD 'POCD') | Up to 5 years
  The non-computerized neuropsychological trail making test is used as an indicator screening test for relevant cognitive changes after the operation. The cut-off is an increase in TMT-B test performance of> 55 seconds three and / or 12 months after the operation compared to the baseline value.
Findings from outpatient neurocognitive evaluation (memory clinic) | Up to 1 year
  Results from patient neurocognitive assessment in a memory clinic are evaluated.
Neuroimaging | Up to 5 years
  Technique to image the nervous system.
Normative database | Up to 5 years
  Establishment of a norm database for deriving normative data in a cooperation between the Clinial Research Unit Berlin/Institute of Health (BIH), the Department of Anesthesiology and Operative Intensive Care Medicine (CCM/CVK) at Charité Universitätsmedizin Berlin and Cambridge Cognition.
Perioperative cognitive disorders | Up to 5 years
  Perioperative cognitive disorders for different surgical cohorts are evaluated to describe domain-specific changes over time in formal cognitive tests. These analyzes are carried out in a joint evaluation with Monument Therapeutics as part of a cooperation agreement
Computerized cognitive data | Up to 5 years
  Computerized cognitive data from CANTAB-research suite, CANTAB eclipse and CANTAB connect
Paper-based, non-computerized, cognitive test data | Up to 5 years
  Paper-based, non-computerized, cognitive test data are data from such as IQ equivalent (e.g. MWT-A), MMSE, MOCA, MMQ, Mini-Cog, etc.
Socio-economic Information 1 | Up to 5 years
  Soci-economic information is collected by FIMA
Socio-economic Information 2 | Up to 5 years
  Soci-economic information is collected by a questionnaire according to Nikolaus 1. Subscale
Comorbidities | Up to 5 years
  Comorbidities are new diagnoses from hospital records.
Charlson comorbidity index | Up to 5 years
  Comorbidity scores
Lifestyle Risks 1 | Up to 5 years
  Consumption of alcohol per week.
Lifestyle Risks 2 | Up to 5 years
  Consumption of tobacco and nicotine is measured by Fagerström Test for Cigarette Dependence (FTCD). Questionnaire scored 0-10 points with Total Score equal to the sum of all points
Level of education | Up to 5 years
  Level of education is measured by ISCED
Incidence of postoperative delirium | Up to 5 years
  Incidence of postoperative delirium is measured by DDS, DSM-V, CAM/CAM-ICU, NuDESC and Chart review
Duration of postoperative delirium | Up to 5 years
  The Duration of postoperative Delirium is measured in days
Severity of postoperative delirium 1 | Up to 5 years
  Severity of delirium 1 is measured by Delirium Detection Score (DDS). The DDS is composed of eight criteria (orientation, hallucination, agitation, anxiety, seizures, tremor, paroxysmal sweating, and altered sleep- wake rhythm). Each item is cored 0,1,4, or 7 points for a possible total score of 0 to 56). Positive if >7.
Severity of postoperative delirium 2 | Up to 5 years
  Severity of delirium 2 is measured by Confusion assessment method-short (CAM-S). This is a CAM-based scoring system for delirium severity. The CAM-S uses the same items as the original CAM and rates each symptom 0 for absent, 1 for mild, or 2 for marked; acute onset of fluctuation receives 0 (absent) or 1 (present) (scored 0-10, higher worse).
Severity of postoperative delirium 3 | Up to 5 years
  Severity of delirium 3 is measured by DSR-R-98. DRS-R-98 is 16 items clinician rated scale. Total Item: 16 = 3 (for diagnosis) + 13 (for severity).
Severity of postoperative delirium 4 | Up to 5 years
  Severity of delirium 4 is measured by ICDSC. Give a score of "1" to each of the 8 items below if the patient clearly meets the criteria defined in the scoring instructions. Give a score of "0" if there is no manifestation orunable to score. If the patient scores >4, notify the physician. The diagnosis of delirium is made following clinical assessment. assessment.
Severity of postoperative delirium 5 | Up to 5 years
  Severity of delirium 5 is measured by Nursing Delirium Screening Scale (Nu-DESC). The Nu-DESC is a scale that evaluates the severity of the 5 delirium characteristics on a scale of 0 (not present) to 2 (severe) and takes only 1-2 min to complete, based on the nurses' observations of the patient's behavior during their shifts.
Length of hospital stay | Up to 5 years
  Participants will be followed for the duration of hospital stay, an expected average of 7 days
Quality of life - relatives | Up to 5 years
  Quality of life is measured by CarerQoL
Quality of life - self 1 | Up to 5 years
  Quality of life is measured by EQ-5D.An index calculated from the five EQ-5D (3L and 5L) dimensions by attaching specific weights to each severity level in each dimension.
Quality of life - self 2 | Up to 5 years
  Quality of life is measured by WHO-5. WHO-5 is a short and generic global rating scale measuring subjective well-being, the respondent is asked to rate how well each of the 5 statements applies to him or her when considering the last 14 days. Each of the 5 items is scored from 5 (all of the time) to 0 (none of the time). The raw score ranges from 0 (absence of well-being) to 25 (maximal well-being). Scores are then converted to a percentage scale from 0 (absent) to 100 (maximal). Higher scores represent greater psychological well-being.
Functional impairment (IADL) 1 | Up to 5 years
  Instrumental Activities of Daily Living (IADLs) < 8
Functional impairment (ADL) 2 | Up to 5 years
  Activities of Daily Living (ADLs) < 100
Depression 1 | Up to 5 years
  Depression 1 is measured by PHQ-8
Depression 2 | Up to 5 years
  Depression 2 is measured by GDS
Anxiety scales | Up to 5 years
  Anxiety is measured by GAD-7
Pain | Up to 5 years
  Pain is measured by different scales, e.g. Numeric Rating Scale
Depth of sedation | Up to 5 years
  The sedation is emasured intraoperatively processed electroencephalogram (EEG) Full-brain EEG recording with surface electrodes, raw EEG analysis measured during the operation.
Sedation | Up to 5 years
  Sedation is measured by the Richmond Agitation Sedation Scale
Type of operation | Up to 5 years
  Type of operation is measured by OPS-Code.
Type of anesthesia | Up to 5 years
  There are four main categories of anesthesia used during surgery and other procedures: general anesthesia, regional anesthesia, sedation (sometimes called "monitored anesthesia care"), and local anesthesia.
Type of concomitant medication | Up to 5 years
  The medication administered during the hospital stay is documented.
Anticholinergic Load | Up to 5 years
  Measured by anticholinergic drug scale
Frailty | Up to 5 years
  Frailty is measured with a modified frailty score according to Fried´s frailty phenotype assessment.
Number of participants with changes in laboratory values 1 | Up to 5 years
  Laboratory results in the hospital including hemoglobin, lymphocytes, total neutrophils, platelet count, white blood cell (WBC) count and inflammatory markers from blood samples.
Number of participants with changes in laboratory values 2 | Up to 5 years
  Laboratory results in the hospital from serum samples
Number of participants with changes in laboratory values 3 | Up to 5 years
  Laboratory results in the hospital from urine samples
Number of participants with changes in laboratory values 4 | Up to 5 years
  Laboratory results in the hospital from stool samples
Perioperative Electroencephalography | During hospital stay an expected avarage of 7 days
  Electroencephalography (EEG)- Mapping with electrodes.
Nutritional status 1 | Up to five years
  Nutritional status 1 is measured by calf circumference
Nutritional status 2 | Up to five years
  Nutritional status 2 is measured by arm circumference
Nutritional status 3 | Up to five years
  Nutritional status 3 is measured by changes in weight
Nutritional status 4 | Up to five years
  Nutritional status 4 is measured by changes in body mass index
Nutritional status 5 | Up to five years
  Nutritional status 5 is measured by questions regarding microbiome
Nutritional status 6 | Up to five years
  Nutritional status 6 is measured by Medi-Score
Nutritional status 7 | Up to five years
  Nutritional status 7 is measured by MNA-SF
Nutritional status 8 | Up to five years
  Nutritional status 8 is measured by Sarcopenia, which is identified by criterion 1: low muscle strength, criterion 2: low muscle quantity and criterion 3: low physical performance. Probable sarcopenia is identified by Criterion 1. Diagnosis is confirmed by additional documentation of Criterion 2.
  If Criteria 1, 2 and 3 are all met, sarcopenia is considered severe.
Inhospital diet | Up to five years
  Inhospital diet is measured by patient record.
Eating habits | Up to five years
  Eating habits are measured by patient survey.

OTHER OUTCOMES:
Demographics | Up to 5 years
  Demographics are measured by demographic data.
Neurological diseases | Up to 5 years
  Neurological diseases are taken from the hospital record
Waist circumference | Up to 5 years
  Waist circumference is measured in cm.
Hip circumfernece | Up to 5 years
  Hip circumference is measured in cm.
Obesitas | Up to 5 years
  Obesitas is measured by body mass index.
Metamemory Questionnaire (MMQ) contentment scale | At Baseline
  Metamemory Questionnaire (MMQ) contentment scale is a participant-reported measure of memory satisfaction, ability, and strategy use..
Presurgical Cognitive Impairment (PreCI) | At Baseline
  Presurgical cognitive impairment is determined as cognitive performance of a test battery.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Charite University, Berlin, Germany
Locations (2):
- Germany (2):
  - Irmgard Landgraf, Berlin
  - Department of Anesthesiology and Operative Intensive Care Medicine Berlin (CCM, CVK), Charité - Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasmussen LS, Larsen K, Houx P, Skovgaard LT, Hanning CD, Moller JT; ISPOCD group. The International Study of Postoperative Cognitive Dysfunction. The assessment of postoperative cognitive function. Acta Anaesthesiol Scand. 2001 Mar;45(3):275-89. doi: 10.1034/j.1399-6576.2001.045003275.x. PMID 11207462
- [Background] Evered L, Silbert B, Knopman DS, Scott DA, DeKosky ST, Rasmussen LS, Oh ES, Crosby G, Berger M, Eckenhoff RG; Nomenclature Consensus Working Group. Recommendations for the nomenclature of cognitive change associated with anaesthesia and surgery-2018. Br J Anaesth. 2018 Nov;121(5):1005-1012. doi: 10.1016/j.bja.2017.11.087. Epub 2018 Jun 15. PMID 30336844